CLINICAL TRIAL: NCT00980369
Title: Incision Type for Lateral Internal Sphincterotomy
Brief Title: The Importance of Lateral Internal Sphincterotomy Incision: Parallel or Vertical
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Feyzullah Ersoz - Serkan Sarı, Istanbul Education and Research Hospital
Other Study IDs: SBIstanbul; 2. General Surgery
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Anal Fissure
Keywords: Lateral internal sphincterotomy; Anal fissure; Surgical technique; Incision; Wound healing
MeSH Terms: conditions — Fissure in Ano; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic anal fissures: Group A: with vertical incision Group B: with parallel incision
- Parallel incision, vertical insicion

SUMMARY:
The purpose of this study is to determine effective incision type for the treatment of chronic anal fissures.

DETAILED DESCRIPTION:
The lateral internal sphincterotomy (LIS) technique is considered the optimal surgical treatment for chronic anal fissures (CAFs); however, questions remain regarding the best technique. The present study investigated whether the type of anoderm incision (vertical or parallel to the anus) affected wound healing, wound-related complications, incontinence and recurrence rates in CAF patients undergoing open LIS.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open lateral internal sphincterotomy for chronic anal fissure

Exclusion Criteria:

* Younger than 18 and older than 65 years of age, patients who had undergone no previous medical treatment, patients with a history of perianal interventions, patients with inflammatory bowel disease, diabetic patients, patients on steroids and immunosuppressives, patients with collagen tissue diseases, mentally retarded patients and patients with malignant disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Estimated); Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Feyzullah Ersoz, Study Chair — Istanbul Education and Research Hospital, General surgery clinic
Locations (1):
- SB Istanbul Education and Research Hospital, Istanbul, Turkey (Türkiye)